CLINICAL TRIAL: NCT07395154
Title: COMPARATIVE EFFECT OF INTEGRATED NEUROMUSCULAR INHIBITION TECHNIQUE AND ACTIVE RELEASE TECHNIQUE ON PAIN, RANGE OF MOTION AND FUNCTIONAL DISABILITY IN PATIENTS WITH UPPER TRAPEZIUS TRIGGER POINTS
Brief Title: Comparison of Integrated Neuromuscular Inhibition Technique (INIT) and Active Release Technique (ART) in Patients With Upper Trapezius Trigger Points
Acronym: INIT ART
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UBAS/ERB/FoRS/25/023
Record Dates: First submitted 2025-12-01; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Myofascial Pain Syndrome
Keywords: Integrated Neuromuscular Inhibition Technique; Active Release Technique; Muscle Energy Technique; Ischemic Compression
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Integrated Neuromuscular Inhibition Technique
  Interventions: Other: Group A
- Group B (Experimental): Active Release Technique
  Interventions: Other: Group B

INTERVENTIONS:
Other: Group A — Participants will receive treatment three times per week for 6 weeks. Each session will begin with a moist hot pack for 10 minutes followed by TENS for 15 minutes to relax the muscles and reduce pain. After this preparation, participants will receive 15 minutes of Integrated Neuromuscular Inhibition Technique, including ischemic compression, strain-counterstrain, and muscle energy technique, applied to the identified myofascial trigger points.
  Other Names: Integrated Neuromuscular Inhibition Technique
  Arms: Group A
Other: Group B — Participants will receive treatment three times per week for 6 weeks. Each session will begin with a moist hot pack for 10 minutes and TENS for 15 minutes to prepare the tissues. This will be followed by 15 minutes of Active Release Technique, including repeated active passes, targeted fiber release, and mild stretching, applied to the upper trapezius myofascial trigger points.
  Other Names: Active Release Technique
  Arms: Group B

SUMMARY:
The goal of this clinical trial is to determine whether two manual therapy techniques-Integrated Neuromuscular Inhibition Technique (INIT) and Active Release Technique (ART)-can reduce pain, improve neck range of motion, and decrease functional disability in adults with upper trapezius myofascial trigger points.

The main questions it aims to answer are:

Does INIT reduce pain, improve ROM, and reduce functional disability more effectively than ART?

Does ART provide similar or different treatment benefits compared to INIT?

Researchers will compare INIT with ART to see which technique produces greater improvements in pain, ROM, and functional disability.

Participants will:

Receive treatment sessions of either INIT or ART.

Undergo assessment of pain, cervical range of motion, and functional disability before and after the intervention.

DETAILED DESCRIPTION:
Myofascial trigger points in the upper trapezius are a common cause of neck pain, restricted cervical mobility, and functional limitations. Manual therapy techniques are frequently used to deactivate trigger points and improve muscle function, but evidence comparing specific techniques remains limited.

This study investigates two commonly used interventions: the Integrated Neuromuscular Inhibition Technique (INIT), which combines sustained pressure, muscle energy technique, and stretching; and the Active Release Technique (ART), which involves movement-based soft tissue release. Both techniques target trigger point sensitivity and muscle tightness but use different mechanisms.

Participants with diagnosed upper trapezius trigger points will be randomly assigned to receive either INIT or ART. Each group will follow a structured treatment protocol over a defined period. Pain intensity, cervical range of motion, and functional disability will be measured at baseline and after the intervention using validated outcome tools.

The study aims to provide comparative evidence on which technique offers greater clinical effectiveness for reducing pain, improving cervical mobility, and enhancing function in individuals with upper trapezius trigger points. Results may assist clinicians in selecting more effective manual therapy strategies for managing myofascial pain.

ELIGIBILITY:
Inclusion Criteria:

* Presence of active trigger points in the upper trapezius muscle.
* Forward Head Posture (measured by craniovertebral angle).
* Pain duration less than 3 months.

Exclusion Criteria:

* History of trauma or surgery involving the cervical spine or shoulder
* Neurological disorders (e.g., cervical radiculopathy)
* Systemic conditions like diabetes or rheumatoid arthritis
* Use of corticosteroids
* Fibromyalgia, Thoracic Outlet Syndrome, Temporomandibular Joint Disorders

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Goniometer (Range of Motion) | Assessment at baseline, after 3rd and 6th weeks.
  The Universal Goniometer (UG) will be used to assess Active Cervical Range of Motion (ACROM) in multiple planes. This reliable tool allows physical therapists to measure joint angles accurately, both with and without assistance. In this study, it will be employed to evaluate cervical spine movement as an objective outcome measure of participants' range of motion.
Numeric Pain Rating Scale (NPRS) | Assessment at baseline, after 3rd and 6th weeks.
  The NPRS questionnaire is composed of an 11-point scale from 0 to 10. The patient chooses the most compatible value for the force of pain they have experienced in the last 24 h, with "0" meaning no pain and "10" meaning intense pain. The patient has to mark the score on the questionnaire according to the pain intensity he/she is experiencing.
Neck Disability Index (NDI) | Assessment at baseline, after 3rd and 6th weeks.
  The Neck Disability Index (NDI) is a ten-item questionnaire that assesses disability associated with neck pain and whiplash. There are four items that relate to subjective symptomatology (pain intensity, headache, concentration, and sleeping) and six items that relate to activities of daily living (lifting, work, driving, recreation, personal care, and reading). The questionnaire requires only 5-10 minutes to complete and score, and requires no special training to administer.

REFERENCES:
- [Background] Sadria G, Hosseini M, Rezasoltani A, Bagheban AA, Davari A, Seifolahi AJJob, et al. A comparison of the effect of the active release and muscle energy techniques on the latent trigger points of the upper trapezius. 2017;21(4):920-5.
- [Background] Nayak PP. A Study to Find Out the Efficacy of Init (Integrated Neuromuscular Inhibition Technique) with Therapeutic Ultrasound Vs Init with Placebo Ultrasound in the Treatment of Acute Myofascial Trigger Point in Upper Trapezius: Rajiv Gandhi University of Health Sciences (India); 2013.
- See also: Related Info — https://search.proquest.com/openview/f0d62b03fcfbe9404ce67fe715b17b2e/1?pq-origsite=gscholar&cbl=2026366&diss=y